CLINICAL TRIAL: NCT04912791
Title: A National Survey on Obstetric Anesthesia and Analgesia Care: Obstetric Anaesthesia And Analgesia Month Attributes - in COVID-19 (OBAAMA-COV)
Brief Title: Obstetric Anaesthesia And Analgesia Month Attributes - in COVID-19
Acronym: OBAAMA-COV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other); Institute of Biostatistics and Analyses, Masaryk University Brno (Unknown); Czech Society of Anaesthesiology, resuscitation and intensive care (ČSARIM) (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: MU_IBA2021
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Obstetric Anesthesia Care
Keywords: Obstetric anesthesia; Survey; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Anesthesia, Obstetrical; Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women in labor undergoing anesthesia care: Women in labor undergoing anesthesia care
  Interventions: Procedure: Obstetric anesthesia and analgesia

INTERVENTIONS:
Procedure: Obstetric anesthesia and analgesia — All anesthesia procedures during labor: labor analgesia, anesthesia for Cesarean section, anesthesia for procedures in third stage of labor

SUMMARY:
A national survey of current practices, preferred drug and technique choices for obstetric anesthesia and analgesia and to evaluate the impact of COVID-19 pandemic on obstetric anesthesia and analgesia in Czech Republic and Slovak Republic

DETAILED DESCRIPTION:
A one month-long project monitoring an obstetric anesthesia practices in obstetric/anesthesia departments throughout the Czech Republic and Slovak Republic.

Electronic Case Report Form (eCRF) is used to collect data on all obstetric anesthesia procedures in peripartal period and obstetric and anesthesia complications. All consecutive cases in each participating center during the study period are recorded. Each record is related to parturient and contains the following sections: history, form of labour analgesia, type of anesthesia for Cesarean section and anesthesia in third stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Women in labor undergoing anesthesia care

Exclusion Criteria:

* not meeting inclusion criteria

Ages: 16 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women in labor
Study Population: Women in labor undergoing anesthesia care
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
A national survey of current practice of obstetric anesthesia and analgesia in Czech Republic and Slovak Republic | Parturition period, up to 24 hours after labor
  Monitoring of all obstetric anesthesia procedures in peripartal period and anesthesia complications: history, form of labour analgesia, type of anesthesia for Cesarean section and anesthesia in third stage of labor.

SECONDARY OUTCOMES:
Types of anesthesia a analgesia in peripartal period | Parturition period, up to 24 hours after labor
  To describe current practice related to peripartal anesthesia care
Complications related to obstetric anesthesia care | Parturition period, up to 24 hours after labor
  To describe current practice a complications related to peripartal anesthesia care

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., Study Chair — University Hospital Brno
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided